CLINICAL TRIAL: NCT02555098
Title: A Bilateral Dispensing Clinical Trial of Sapphire Lens Against Senofilcon A Toric for Astigmatism Lens Over 2 Weeks
Brief Title: A Bilateral Dispensing Clinical Trial of an Sapphire Lens Against Senofilcon A Toric for Astigmatism Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CV-15-15
Record Dates: First submitted 2015-09-04; First posted 2015-09-21 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sapphire contact lenses (Experimental): Each subject randomized to wear either the Investigational lenses (test) or senofilcon A contact lenses (control) as a matched pair and cross over to the second matched pair.
  Interventions: Device: Sapphire contact lenses
- senofilcon A (Active Comparator): Each subject randomized to wear either the Investigational lenses (test) or senofilcon A contact lenses (control) as a matched pair and cross over to the second matched pair.
  Interventions: Device: senofilcon A contact lenses

INTERVENTIONS:
Device: Sapphire contact lenses — Each subject randomized to wear either the test or control contact lenses as a matched pair and cross over to the second matched pair
  Arms: Sapphire contact lenses
Device: senofilcon A contact lenses — Each subject randomized to wear either the test or control contact lenses as a matched pair and cross over to the second matched pair
  Arms: senofilcon A

SUMMARY:
This study was conducted to evaluate the clinical performance of an investigational silicone-hydrogel lens against Senofilcon A toric lens.

The study results were not used for design validation of the investigational product.

DETAILED DESCRIPTION:
This will be a randomized, bilateral, 2-week cross-over, double-masked, dispensing study comparing the investigational test lens against the Senofilcon A Toric for Astigmatism control lens.

ELIGIBILITY:
Inclusion Criteria:

* A person is eligible for inclusion in the study if they:

  1. Are at least 18 years of age and have full legal capacity to volunteer;
  2. Have read and signed an information consent letter;
  3. Are willing and able to follow instructions and maintain the appointment schedule;
  4. Are an adapted soft contact lens wearer;
  5. Require spectacle lens powers in both eyes;

     1. Sphere: between -1.75 to -6.00 diopters and
     2. Astigmatism: between -1.00 to -2.25 and
     3. Axis: 180 ± 20 degrees
  6. Are willing to wear contact lenses in both eyes;
  7. Have manifest refraction visual acuities (VA) equal to or better than logMAR (log of the minimum angle of resolution) equivalent of 20/25 in each eye;
  8. To be eligible for lens dispensing, the subject must have VA of logMAR equivalent of 20/30 or better in each eye with the study lenses and the investigator must judge the fit including toric orientation as acceptable.

Exclusion Criteria:

* A person will be excluded from the study if they:

  1. Are participating in any concurrent clinical or research study;
  2. Have any known active* ocular disease and/or infection;
  3. Have a systemic condition that in the opinion of the investigator may affect a study outcome variable;
  4. Are using any systemic or topical medications that in the opinion of the investigator may affect a study outcome variable;
  5. Have known sensitivity to the diagnostic pharmaceuticals to be used in the study;
  6. Are pregnant, lactating or planning a pregnancy at the time of enrolment (by verbal confirmation at the screening visit);
  7. Are aphakic;
  8. Have undergone refractive error surgery;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michel Guillon, Principal Investigator — Ocular Technology Group
Locations (1):
- Family Eye Care Center, Campbell, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sapphire Test Lenses Then Senofilcon A Lenes: Each subject was randomized to wear the Investigational lenses (test) for two weeks then cross-over to senofilcon A contact lenses (control) for two weeks.
  Sapphire contact lenses: Contact Lenses Senofilcon A : Contact lenses
- Senofilcon A Then Sapphire Test Lenses: Each subject was randomized to wear the senofilcon A contact lenses (control) for two weeks then cross-over to Sapphire lenses (test) for two weeks.
  Senofilcon A : Contact lenses Sapphire lenses: Contact Lenses
Period: First Intervention
Arm/Group | Sapphire Test Lenses Then Senofilcon A Lenes | Senofilcon A Then Sapphire Test Lenses
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Sapphire Test Lenses Then Senofilcon A Lenes | Senofilcon A Then Sapphire Test Lenses
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Each subject randomized to wear either the Investigational lenses (test) or senofilcon A contact lenses (control) as a matched pair and cross over to the second matched pair.
Groups:
- Overall Study: Each subject randomized to wear either the Sapphire lenses (test) or senofilcon A contact lenses (control) as a matched pair for two weeks and cross over to the second matched pair for two weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Subjective Ratings for Comfort
Description: Scale 0-100; (0=Cannot be worn; 100=Cannot be felt ever)
Time Frame: Baseline (10 minutes post lens settling)
Population: One subject was excluded from the analysis due to compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sapphire Lenses: Each subject randomized to wear the Sapphire lenses (test) for two weeks.
  Sapphire lenses: Contact lenses
- Senofilcon A: Each subject randomized to wear senofilcon A contact lenses (control) for two weeks.
  senofilcon A contact lenses: Contact lenses
Arm/Group | Sapphire Lenses | Senofilcon A
Number analyzed (Participants) | 22 | 22
units on a scale | 89 (14) | 80 (20)

2. Primary Outcome: Subjective Ratings for Comfort
Description: Scale 0-100; (0=Cannot be worn; 100=Cannot be felt ever)
Time Frame: 2 weeks
Population: One subject was excluded from the analysis due to compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sapphire Lenses: Each subject randomized to wear the Sapphirel lenses (test) for two weeks.
  Sapphire lenses: Contact lenses
Arm/Group | Sapphire Lenses | Senofilcon A
Number analyzed (Participants) | 22 | 22
units on a scale | 85 (18) | 72 (27)

3. Primary Outcome: Subjective Ratings for Comfort Preference
Description: Subjective Ratings for Comfort Preference: Sapphire lens, senofilcon A lens, No preference
Time Frame: Baseline (10 minutes post lens settling)
Population: One subject was excluded from the analysis due to compliance.
Measure: Number; unit: percentage of participants
Groups:
- Overall Study: Each subject randomized to wear the Sapphire lenses (test) and senofilcon A contact lenses for two weeks in this cross-over study.
  Sapphire contact lenses: Contact lenses senofilcon A contact lenses : Contact lenses
Arm/Group | Overall Study
Number analyzed (Participants) | 22
percentage of participants
  Sapphire lens | 46
  senofilcon A | 18
  No Preference | 36

4. Primary Outcome: Subjective Ratings for Comfort Preference
Description: Subjective Ratings for Comfort Preference: Sapphire lens, senofilcon A lens, No preference
Time Frame: 2 weeks
Population: One subject was excluded from the analysis due to compliance.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 22
percentage of participants
  Sapphire lens | 68
  senofilcon A | 27
  No Preference | 5

5. Primary Outcome: Subjective Assessment of Visual Quality
Description: Subjective assessment of visual quality assessed on a Scale: 0-100 (0=Extremely poor vision all of the time; Cannot function; 100=Excellent vision all of the time)
Time Frame: Baseline (10 minutes post lens settling)
Population: One subject was excluded from the analysis due to compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sapphire Contact Lenses: Each subject randomized to wear the Sapphire lenses (test) for two weeks.
  Sapphire contact lenses: Contact lenses
Arm/Group | Sapphire Contact Lenses | Senofilcon A
Number analyzed (Participants) | 22 | 22
units on a scale | 85 (15) | 85 (21)

6. Primary Outcome: Subjective Assessment of Visual Quality
Description: as for outcome 5
Time Frame: 2 weeks
Population: One subject was excluded from the analysis due to compliance.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire Contact Lenses | Senofilcon A
Number analyzed (Participants) | 22 | 22
units on a scale | 81 (19) | 73 (27)

7. Primary Outcome: Subjective Assessment of Overall Satisfaction
Description: Subjective assessment of overall satisfaction on a Scale: 0-100: (0=Extremely dissatisfied; 100=Extremely satisfied)
Time Frame: Baseline (10 minutes post lens settling)
Population: One subject was excluded from the analysis due to compliance
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Sapphire Lenses: Each subject randomized to wear the Sapphire lenses (test) for two weeks.
  Sapphire contact lenses: Contact lenses
Arm/Group | Sapphire Lenses | Senofilcon A
Number analyzed (Participants) | 22 | 22
units on a scale | 89 (12) | 81 (21)

8. Primary Outcome: Subjective Assessment of Overall Satisfaction
Description: Subjective assessment of overall satisfaction on a Scale: 0-100: (0=Extremely dissatisfied; 100=Extremely satisfied)
Time Frame: 2 weeks
Population: One subject was excluded from the analysis due to compliance
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sapphire Contact Lenses | Senofilcon A
Number analyzed (Participants) | 22 | 22
units on a scale | 87 (14) | 73 (30)

9. Primary Outcome: Subjective Overall Preference
Description: Subjective Overall Preference: Sapphire lens, senofilcon A lens, No preference
Time Frame: Baseline (10 minutes post lens settling)
Population: One subject was excluded from the analysis due to compliance.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 22
percentage of participants
  Sapphire Lens | 55
  No Preference | 18
  senofilcon A | 27

10. Primary Outcome: Subjective Overall Preference
Description: Subjective Overall Preference: Sapphire lens, senofilcon A lens, No preference
Time Frame: 2 weeks
Population: One subject was excluded from the analysis due to compliance.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Study
Number analyzed (Participants) | 22
percentage of participants
  Sapphire Lens | 73
  No Preference | 4
  senofilcon A | 23

ADVERSE EVENTS:
Time Frame: From dispense up to 2 weeks on each study lenses, a total of 4 weeks.
Arm/Group | Sapphire Contact Lenses | Senofilcon A
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No